CLINICAL TRIAL: NCT07354542
Title: Comparison of the Effects of Virtual Reality-based and Traditional Relaxation Therapy on Postoperative Pain and Sleep Quality in Patients Undergoing Hip and Knee Replacement Surgery
Brief Title: Effects of Different Relaxation Therapies on Pain and Sleep in Hip and Knee Arthroplasty Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Meltem Soydan, Nurse, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BartınU-SBF-MS-01
Record Dates: First submitted 2025-12-23; First posted 2026-01-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis (OA) of the Hip; Osteoarthritis (OA) of the Knee
Keywords: Postoperative Pain; Sleep Quality; Virtual Reality
MeSH Terms: conditions — Osteoarthritis; Pain, Postoperative; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality-Based Relaxation Group (Experimental): Participants receive relaxation exercises delivered through virtual reality technology following hip and knee replacement surgery. The intervention is provided during the postoperative period in addition to standard care.
  Interventions: Behavioral: Virtual Reality-Based Relaxation
- Traditional Relaxation Therapy Group (Active Comparator): Participants receive traditional relaxation exercises without virtual reality following hip and knee replacement surgery. The intervention is provided during the postoperative period in addition to standard care.
  Interventions: Behavioral: Traditional Relaxation Therapy

INTERVENTIONS:
Behavioral: Virtual Reality-Based Relaxation — Relaxation exercises delivered through virtual reality technology during the postoperative period following hip and knee replacement surgery.
  Arms: Virtual Reality-Based Relaxation Group
Behavioral: Traditional Relaxation Therapy — Standard relaxation exercises performed without virtual reality during the postoperative period following hip and knee replacement surgery.
  Arms: Traditional Relaxation Therapy Group

SUMMARY:
Hip and knee replacement surgery is commonly performed in older adults. After surgery, many patients experience pain, limited movement, and sleep problems. These difficulties can make daily activities such as walking or climbing stairs more challenging and may reduce quality of life during recovery.

Relaxation exercises are often used to help reduce pain and improve sleep after surgery. Virtual reality (VR) is a technology that provides a multisensory experience and may help people relax by shifting their attention away from pain and discomfort.

This study is designed to compare two different relaxation approaches used after hip and knee replacement surgery. One group of patients will perform relaxation exercises using virtual reality, while another group will perform traditional relaxation exercises. The study will examine pain levels and sleep quality in both groups.

The results of this study may help to better understand whether virtual reality-based relaxation can be used as an alternative or supportive method for managing pain and sleep problems after joint replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Those who volunteered to participate in the research,
* 18 years and older,
* No diagnosed mental or sleep problems, epilepsy, or depression,
* No vision, hearing, or speech problems,
* Those who speak Turkish,
* Knee and hip replacement surgery ,
* No active nausea or vomiting prior to the virtual reality application,
* According to the Numerical Rating Scale, the patient reports pain.
* Those receiving analgesia treatment according to clinical protocol,
* Anyone who owns a mobile phone or tablet capable of playing videos, using any brand of internet provider,
* Patients who had not previously practiced breathing exercises were included .

Exclusion Criteria:

* Having a problem that prevents communication,
* Being admitted to the ward where the surgery and study were performed at another center,

  . Complications develop after knee and hip replacement surgery,
* Nausea and vomiting may occur during the procedure.
* Wanting to withdraw from the research,
* Experiencing chronic pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | Postoperative three days period
  Pain intensity will be assessed using Numerical Rating Scale (0-10 points) in patients undergoing hip and knee replacement surgery. 0 represents no pain and 10 represents the most severe pain.

SECONDARY OUTCOMES:
Sleep Quality | Postoperative three days period
  Sleep quality will be evaluated using Richards Campbell Sleep Questionnaire (0-100 points) during the postoperative period.The scale uses a score range of "0-25" to indicate very poor sleep and a score range of "76-100" to indicate very good sleep. The total score is evaluated based on 5 items; item 6, which assesses the noise level in the environment, is excluded from the total score evaluation. As the score obtained from the questionnaire increases, it is interpreted that the patients' sleep quality has improved.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Çelik, Professor, Study Director — Bartin University Health Science Faculty
Locations (1):
- Bartın State Hospital, Bartın, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No